CLINICAL TRIAL: NCT03506659
Title: Electrochemical Skin Conductance in Evaluation of Chronic Neuropathy
Brief Title: Electrochemical Skin Conductance in Evaluation of Chronic Neuropathy électrochimique cutanée
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion rate too low
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SUDOKU
Record Dates: First submitted 2018-03-15; First posted 2018-04-24 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Difference, Individual

STUDY DESIGN:
Intervention Model Description: Parallel group open label Monocentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Active Comparator): 2000 patients healthy in anesthesiology consultation
  Interventions: Device: SUDO-SCAN Device
- Patients (Experimental): 2000 patients in pain clinic consultation
  Interventions: Device: SUDO-SCAN Device

INTERVENTIONS:
Device: SUDO-SCAN Device — Sudo-scan is a machine with 2 palets for hands and 2 palets for foots. The patient has to put his 2 hands and 2 foots on the machine. The machine do the measures during 2 minutes.

SUMMARY:
Use of cutaneous electrochemical conductance for preclinical screening of small-caliber nerve fibers

DETAILED DESCRIPTION:
Objective: Use of cutaneous electrochemical conductance for preclinical screening of small-caliber nerve fibers

Background:

Sudoscan is a tool developed to evaluate and screen peripheral neuropathies in diabetes. His indication has been extended to other neuropathies such as post-chemotherapy, Fabry's disease, Parkinson's disease, familial amyloid polyneuropathy.

Main objective: Evaluation of the relevance of cutaneous electrochemical conductance in chronic peripheral neuropathies.

Methodology :

Recruitment of 2 groups of 2000 patients Group 1: Patients with chronic neuropathy, during clinic bread consultation Group 2: Patients to benefit from scheduled surgery seen during anesthesia consultation For both groups filling the central awareness inventory questionnaire

Analysis of the results after the recruitment has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult

Exclusion Criteria:

* Patients group : Not have a chronic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Difference of timing for Electrochemical skin conductance | 3 minutes
  the investigators will measure the timing between the 4 members for the Electrochemical skin conductance

CONTACTS AND LOCATIONS:
Overall Officials: Turgay TUNA, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- ERASME Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided